CLINICAL TRIAL: NCT01802112
Title: Randomised Controlled Trial of Efficacy of Resistant Maltodextrins on Reducing Colonic Transit Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Antonio Technologies - San Antonio Catholic University of Murcia (Other)
Collaborators: Universidad Católica San Antonio de Murcia (Other); Hospital Virgen de la Vega (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROT-001
Record Dates: First submitted 2013-02-22; First posted 2013-03-01 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Constipation
Keywords: Colonic transit; Dietary Fiber; Radiopaque marker
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maltodextrins (Placebo Comparator): 15 grams of maltodextrins per day dissolved in water during 21 days
  Interventions: Other: placebo
- Resistant maltodextrins (Experimental): 15 grams of resistant maltodextrins per day, dissolved in water during 21 days
  Interventions: Dietary Supplement: Resistant maltodextrins

INTERVENTIONS:
Dietary Supplement: Resistant maltodextrins — 15 grams of Resistant maltodextrins per day dissolved in water during 21 days
  Other Names: Fibersol®
  Arms: Resistant maltodextrins
Other: placebo — 15gr placebo
  Arms: Maltodextrins

SUMMARY:
The purpose of this study is to assess the efficacy of resistant maltodextrins, compared to placebo, in reducing the colonic transit time in healthy subjects.

DETAILED DESCRIPTION:
In the last fifty years we have drastically changed our eating habits, in particular our fibre intake. Our hunter-gatherer ancestors ate more than 100 species of fruit and vegetables, which contributed between 20 and 30 g of dietary fibre per day. Currently, a typical citizen of our country reaches 10% of that amount.

Therefore, fibre deficiency alters digestion and metabolism, increasing nutrient absorption (obesity, increased insulin resistance, hyperlipidaemias), produces altered colonic metabolism (inflammatory bowel disease), and slows faecal transit (increasing the lumen pressure with diverticulosis, appendicitis, haemorrhoids and colon cancer. In addition, the prebiotic effect is important.

Several studies have demonstrated the effectiveness of digestion-resistant maltodextrin in the treatment of chronic idiopathic constipation. Investigators carried out a single blind study among young people with constipation who were administered 9.2 grams of resistant maltodextrins per day or placebo, and found significant changes in defecation frequency and in faecal volume.

Kimura et al. carried out a clinical trial in women with constipation and a defecation frequency of less than 3 times per week and administered 5 grams of resistant maltodextrins per day, demonstrating its effectiveness in significantly increasing the number of defecations per week, the number of days per week without defecation and the faecal volume. Additionally, an improvement was found aspects such as colour, stool odour and psychological feeling after defecation.

Finally, an interesting feature of Resistant maltodextrins is that it normalises the colonic transit time without causing diarrhoea, whilst increasing the stool volume, moisture and frequency of defecation.

The purpose of this study is to assess the efficacy of resistant maltodextrins, compared to placebo, in reducing the colonic transit time in healthy subjects.

For That, 60 subjects will be stratified by gender (30 women: 15 with resistant maltodextrins and 15 placebo and 30 men: 15 with resistant maltodextrins and 15 placebo).

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes (men and women) between 18 and 30 years old of Caucasian race selected from the general population
* Subjects capable of understanding the clinical study, willing to provide written informed consent and to fulfil the procedures and requirements of the study.

Exclusion Criteria:

* Diagnosis of a BMI ≥ 30 Kg/m2.
* Individuals with a daily defecation habit.
* Subjects with a history of any digestive disease or who have undergone gastrointestinal surgery (excluding appendicectomy or herniorrhaphy), abdominal surgery in the last two years or any recent major extra-abdominal surgery.
* Subjects with diabetes, hypothyroidism or hyperthyroidism.
* Subjects with a history of systemic disease that might effect gut motility.
* Subjects on dietary treatment and/or drugs that effect body weight or appetite.
* Individuals that have had any change in dietary habit in the last 2 months.
* Subjects with a history of drug or alcohol abuse, or other substances or factors that might limit their ability to cooperate during the study.
* Subjects with bowel habits affected by stress.
* Subjects taking medication or drugs that alter gut motility.
* Pregnant women.
* Subjects that have stopped smoking in the last 6 months or who intend to give up smoking during the study.
* Subjects with allergies or eating disorders.
* Subjects that consume an excessive amount of alcohol (>3 glasses of wine or beer per day)
* Individuals that engage in physical exercise two or more times per week.
* Subjects whose condition makes them ineligible to take part in the study, according to the investigator.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Changes in Colonic Transit Time (CTT) | 28 days from the start of the study
  to determine CTT volunteers should ingest a capsule of radiopaque markers each day for five consecutive days. 24 hours after the final intake of markers an abdominal X-ray should be performed.

SECONDARY OUTCOMES:
Segmental colonic transit time (SCTT) | 28 days from the start of the study
  to determine CTT volunteers should ingest a capsule of radiopaque markers each day for five consecutive days. 24 hours after the final intake of markers an abdominal X-ray should be performed.
Defecation frequency (DF) | 28 days
Stool Consistency | 28 days
  Each of the study subjects will be given a defecation habit diary where consistency of stools from the 28 days of the experimental phase will be recorded according to the Bristol Stool Chart
Stool volume by just their eye observation | 28 days
Clinical Variables of Intestinal Function | 28 days
  these variables will be assessed by determining the number of the Rome III Criteria they fulfil
Assessment of dietary fibre intake | from day 2 to day 6 and from day 23 to day 27
  This outcome will be assessed using a dietary survey. A five-day food record. This food record will be carried out at the same days in both study phases (from day 2 to day 6 and from day 23 to day 27).
  This data will be processed by a computer system that uses internationally validated food composition tables
Efficacy Blood analysis | 28 days
  A blood sample will be taken to determine the blood count and blood biochemistry (glucose, lipid profile, ferritin and ions).
Safety Blood analysis | 29 days
  An analysis of blood biochemistry will be carried out to determine values for enzymes to assess liver function, and biomolecules such as bilirubin, urea and creatinine to assess renal function

OTHER OUTCOMES:
Adverse Events | 29 days
  The safety profile will be assessed using the record of adverse events. Adverse events related to this study will be due to the intake of soluble fibre, the most frequently reported being: flatulence, diarrhoea and gastrointestinal bloating.

CONTACTS AND LOCATIONS:
Locations (1):
- San Antonio Catholic University of Murcia, Guadalupe, Murcia, Spain